CLINICAL TRIAL: NCT04322058
Title: Pathways to Fatherhood and Families: The Dads' Club
Status: Completed | Type: Observational
Sponsor: California State University, San Marcos (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 90FK0105-01-00
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2020-03

CONDITIONS: Fathers

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fathers or paternal caregivers to a child 0-18 years of age: Parenting and Healthy Relationship Education (10 Core 24/7 workshops covering- 15 hours of education), financial and economic mobility programming, comprehensive case management, and supplemental workshops utilizing the Within My Reach curriculum.
  Interventions: Other: The Dads' Club

INTERVENTIONS:
Other: The Dads' Club — The core intervention is Core 24/7 workshop attendance

SUMMARY:
The purpose of this study is to identify changes in parenting, relationship, and financial responsibility outcomes among program participants and to identify processes through which the Dads' Club program affects performance outcomes.

DETAILED DESCRIPTION:
The Dads' Club program services North County San Diego fathers or paternal caregivers to a child 0-18 years of age, speaking English or Spanish, and being willing to attend the program's core parenting workshop.

The program consists of Parenting and Healthy Relationship Education (10 Core 24/7 workshops covering- 15 hours of education), financial and economic mobility programming, comprehensive case management, and supplemental workshops utilizing the Within My Reach curriculum.

Four research questions will be evaluated:

1. What was the magnitude of change in parenting, relationship, and financial responsibility outcomes from program entrance to exit?
2. What was the magnitude of change in parenting, relationship, and financial responsibility outcomes from program entrance to six months post-exit?
3. How was program dose related to change in parenting, relationships, and financial responsibility from program entrance to six months post-exit?
4. How was program support utilization related to change in parenting, relationships, and financial responsibility outcomes from program entrance to exit?

Inclusion in the sample for research questions involving program exit require completion of 80% of the program, defined as completing 8 out of 10 Core 24/7 workshops and a matched pre and post on each question. Inclusion in the sample for research questions involving six month follow-up requires completion of at least 20% of the program, defined as completing two Core 24/7 workshops and a matched pre and post on each question.

ELIGIBILITY:
Inclusion Criteria:

* Father or paternal caregiver of child age 0-18
* Speaks English or Spanish
* Willing to attend program workshops

Exclusion Criteria:

* None

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Fathers or paternal caregivers of child(ren) age 0-18
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Last time saw Child 1 | 1 month
  Father/Child Interaction Measure 1
Reached out Child 1 | 1 month
  Father/Child Interaction Measure 2
Talk to Child 1 | 1 month
  Father/Child Interaction Measure 3
Parenting Practices | 1 month
  University of Idaho Survey of Parenting Practices
Buy Things Child 1 | 1 month
  Financial Responsibility Outcome 1
Pay Bills | 1 month
  Financial Responsibility Outcome 2
Employment Status | 1 month
  Employment Measure 1
Income | 1 month
  Employment Measure 2
Conflict resolution | 1 month
  Satisfaction with partner/spouse conflict resolution

CONTACTS AND LOCATIONS:
Locations (1):
- California State University San Marcos, San Marcos, California, United States

IPD SHARING:
Plan to Share IPD: Undecided